CLINICAL TRIAL: NCT07134335
Title: A Phase II Clinical Study to Evaluate the Efficacy and Safety of UBT251 Injection in Obese/Overweight Chronic Kidney Disease (CKD) Population
Brief Title: UBT251 Injection Phase II Clinical Study (CKD)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The United Bio-Technology (Hengqin) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TUL-UBT251(II-4)202503
Record Dates: First submitted 2025-08-13; First posted 2025-08-21 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-08

CONDITIONS: Obesity &Amp; Overweight; Chronic Kidney Disease
MeSH Terms: conditions — Obesity; Overweight; Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 2.0 mg group (Experimental): Patients will be treated with UBT251 s.c. once weekly for 24 weeks. The starting dose of UBT251 will be 0.5 mg subcutaneous injection with increasing doses at 5, 9 and 13 weeks to 1.0, 2.0 and 2.0 mg once weekly.
  Interventions: Drug: UBT251
- 4.0 mg group (Experimental): Patients will be treated with UBT251 s.c. once weekly for 24 weeks. The starting dose of UBT251 will be 1.0 mg subcutaneous injection with increasing doses at 5, 9 and 13 weeks to 2.0, 4.0 and 4.0 mg once weekly.
  Interventions: Drug: UBT251
- 6.0 mg group (Experimental): Patients will be treated with UBT251 s.c. once weekly for 24 weeks. The starting dose of UBT251 will be 1.0 mg subcutaneous injection with increasing doses at 5, 9 and 13 weeks to 2.0, 4.0 and 6.0 mg once weekly.
  Interventions: Drug: UBT251

INTERVENTIONS:
Drug: UBT251 — Subcutaneous injection once weekly
  Arms: 2.0 mg group
Drug: UBT251 — Subcutaneous injection once weekly
  Arms: 4.0 mg group
Drug: UBT251 — Subcutaneous injection once weekly
  Arms: 6.0 mg group

SUMMARY:
This multicenter, randomized, double-blind, placebo-controlled phase II clinical study to evaluate the efficacy and safety of UBT251 injection in obese/overweight chronic kidney disease (CKD) population

ELIGIBILITY:
Inclusion Criteria:

1. Age 18~75 years old (including border value), BMI >=24 kg/m^2, gender is not limited.
2. Subject estimated glomerular filtration rate (eGFR): >=45 and < 90 mL/min/1.73m^2 (calculated using the CKD-EPI formula).
3. Subjects 300 mg/g <= UACR <= 5000 mg/g 3 months or more prior to screening; At least 2 measurements (not on the same day) within 4 weeks of the screening period, and each measurement must meet this criterion.
4. If treated with SGLT2i, angiotensin-converting enzyme inhibitors (ACEi), angiotensin receptor blockers (ARBs), mineralocorticoid receptor antagonists (MRAs) before screening, a stable dose of >=4 weeks is required unless there are contraindications or intolerance. (For subjects who are intolerant to the above drugs, they can still be included if judged by the investigator to be suitable to participate in the investigator.) )
5. Volunteer to participate in the study and sign the ICF.
6. Female of childbearing potential or male subjects with partners of childbearing potential agree to use effective contraception from the start of study treatment until 3 months after the end of the last dose.

Exclusion Criteria:

1. History or evidence of any of the following diseases: 1) Diagnosis of type 1 diabetes or other special type diabetes. 2) Presence of non-recovered acute kidney injury (AKI) at screening. 3) Previous or current suffering: bilateral renal artery stenosis (stenosis>=50%), tubulointerstitial nephritis, lupus nephritis, autosomal dominant polycystic kidney disease (ADPKD) and autosomal recessive polycystic kidney disease (ARPKD), anti-neutrophil cytoplasmic antibody (ANCA)-associated vasculitis, unilateral nephrectomy or other severe renal structural abnormalities, and a history of unstable or rapidly progressing kidney disease as judged by the investigator. 4) Poorly controlled hypertension (systolic blood pressure >=160 mmHg and/or diastolic blood pressure >=100 mmHg at screening). 5) Glycated hemoglobin (HbA1c) >= 9.5%. 6) Presence of serious illness or medical condition judged by the investigator during the screening period, including but not limited to: a) History of malignant tumor disease within 5 years prior to screening (except for cured basal cell or squamous cell carcinoma of the skin and carcinoma in situ at any site); b) Arterial/venous thrombotic events within 6 months prior to screening, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction [except old lacunar cerebral infarction]), deep vein thrombosis; c) History of internal myocardial infarction or surgery such as percutaneous coronary intervention and coronary artery bypass grafting 6 months before screening; d) History of internal heart failure 6 months prior to screening, with New York Heart Association (NYHA) functional class III. or IV. 7) Combined with gastroparesis or other diseases related to gastrointestinal emptying disorders (such as pyloric obstruction, intestinal obstruction, etc.), uncontrolled gastroesophageal reflux disease, gastrointestinal diseases assessed by the investigator as increasing the risk after medication (such as severe active ulcers, inflammatory bowel disease, acute gastroenteritis, symptomatic chronic gastroenteritis), or undergoing major upper gastrointestinal surgery. 8) History of pancreatitis or pancreatic injury, or pancreatic surgery. 9) History of symptomatic gallbladder disease within 2 years prior to screening, defined as imaging examination suggesting the presence of gallstones and diagnosis-related symptoms related to gallstones; Subjects who have undergone gallstone surgery and/or cholecystectomy (surgery completed at least 3 months prior to screening) with no long-term complications may participate in this study. 10) History or family history of medullary thyroid carcinoma (MTC), multiple endocrine neoplasia (MEN) type 2. 11) History of acute complications of diabetes (diabetic ketoacidosis, diabetic lactic acidosis, hyperglycemic hyperosmolar state, etc.) within 6 months prior to screening. 12) Severe retinal and macular degeneration (including but not limited to proliferative retinopathy, macular edema, retinal detachment, etc.) in the past or at screening, which require further urgent treatment as judged by the investigator. 13) Severe chronic complications of diabetes (including but not limited to severe diabetic neuropathy, diabetic foot, etc.) at screening, and the investigator judges that this complication may affect the compliance and safety of the subjects. 14) Severe hypoglycemia or recurrent symptomatic hypoglycemia within 6 months prior to screening (>=2 times within half a year). 15) Abnormal thyroid function that cannot be controlled with a stable dose of medication, or clinically significant abnormalities in thyroid function test results at screening that require initiation of treatment; 16) History of depression or patient health status questionnaire-9 (PHQ-9) score >=15 points at screening; or a history of severe mental illness (including but not limited to suicidal tendencies or suicide attempts, schizophrenia, bipolar disorder, etc.).
2. Medication history within 3 months prior to randomization that meets any of the following conditions: 1) Receive dipeptidyl peptidase 4 (DPP-4) inhibitors, amylin analogues, glucagon-like peptide-1 (GLP-1) analogues, glucose-dependent insulinic polypeptide (GIP) analogues, glucagon (GCG) analogues. 2) Systemic use of steroid glucocorticoids or immunosuppressants (except for topical or intraarticular, intranasal, and inhaled glucocorticoids; Short-term [<= 7 days] use of glucocorticoids for the prevention or treatment of non-autoimmune allergic diseases). 3) Use of over-the-counter weight loss drugs (including but not limited to orlistat) or food inhibitors (including traditional Chinese medicine), or treatment with lipid-dissolving injections (e.g., lipolysis injections) within 3 months prior to screening.
3. Those who have any of the following test abnormalities during screening: 1) Severe anemia (hemoglobin < 7.0 g/dL); 2) Abnormal liver function (ALT or AST >= 3 ×upper limit of normal [ULN], or serum total bilirubin [TBIL] >= 1.5 × ULN); 3) Serum albumin < 30 g/L; 4) Serum potassium > 5.5 mmol/L; 5) Fasting triglycerides >= 5.6 mmol/L; 6) International normalized ratio (INR) >= 1.5 × ULN; 7) Serum calcitonin level > 50 ng/L; 8) Serum amylase or lipase > 2.0× ULN. 9) Positive hepatitis B surface antigen (HBsAg) test and hepatitis B virus deoxyribonucleic acid (HBV-DNA) higher than the lower limit of detection, positive hepatitis C virus antibody test (HCV-Ab) and hepatitis C virus ribonucleic acid (HCV-RNA) above the upper limit of the reference value range, positive human immunodeficiency virus antibody (HIV-Ab) test at screening, syphilis antibody (TP- Ab) Those who test positive (RPR titer or TRUST test is required, except for cured syphilis). 10) Clinically significant electrocardiogram (ECG) abnormalities at screening (meeting one of them): a) Second or third degree atrioventricular block; b) Long QT syndrome; or QTcF > 470ms for women and > 450ms for males；c) pre-excitation syndrome; d) Other severe arrhythmias requiring treatment; e) Heart rate < 50 beats/min or > 110 beats/min.
4. Body weight change of more than 5% within 6 weeks prior to screening.
5. Those who have had or plan to undergo bariatric surgery during the trial.
6. Those with a history of alcohol and drug abuse.
7. Those who are allergic to the study drug or its excipients.
8. Those who have participated in other clinical trials within 30 days before screening (except for screening only but not medicated or non-interventional studies) or within 5 half-lives of using investigational drugs, whichever is longer.
9. Subject is receiving dialysis/kidney transplantation or plans to undergo dialysis/kidney transplantation during the study.
10. Pregnant or lactating women.
11. Other conditions that the investigator considers unsuitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2030-07-11 (Estimated); Study Completion 2030-07-11 (Estimated)

PRIMARY OUTCOMES:
log-transformed urinary albumin:creatinine ratio（UACR） | 24 weeks
  The change in log-transformed UACR from baseline after 24 weeks of treatment

SECONDARY OUTCOMES:
log-transformed urinary albumin:creatinine ratio (UACR) | 12 weeks
  Change from baseline in log-transformed UACR after 12 weeks of treatment
24-hour urine protein quantification | 12 weeks ，24 weeks
  After 12 weeks and 24 weeks of treatment, the change of 24-hour urine protein quantification from baseline
estimated glomerular filtration rate (eGFR) | 12 weeks，24 weeks
  Change from baseline in eGFR after 12 weeks and 24 weeks of treatment
the proportion of subjects with a reduction of >=30%, >=40%, and >=50% compared with the baseline UACR geometric mean | 12 weeks，24 weeks
  After 12 weeks and 24 weeks of treatment, the proportion of subjects with a reduction of >=30%, >=40%, and >=50% compared with the baseline UACR geometric mean
serum creatinine | 12 weeks，24 weeks
  Change from baseline in serum creatinine after 12 weeks and 24 weeks of treatment
body weight | 12 weeks，24 weeks
  Change in body weight from baseline after 12 weeks and 24 weeks of treatment
EQ-5D-5L score | 24 weeks
  Change from baseline in EQ-5D-5L score after 24 weeks of treatment
EQ-VAS score | 24 weeks
  Change from baseline in EQ-VAS score after 24 weeks of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No